CLINICAL TRIAL: NCT07160413
Title: Peripheral Nerve Activation Sensitivity to Electromagnetic and Electrical Stimulation in the Upper Arm
Brief Title: Peripheral Nerve Activation Sensitivity
Acronym: PERNEAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Niederhauser (Other)
Collaborators: Bern University of Applied Sciences (Other); Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor-Investigator, Thomas Niederhauser, Prof. Dr., Bern University of Applied Sciences
Organization: Bern University of Applied Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-00776; 108.018 IP-LS (Other Grant/Funding Number: Innosuisse)
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Nerve Excitation Sensitivity
Keywords: Peripheral nerve stimulation; Magnetic and electric stimulation; Sensitivity of nerves to magnetic fields

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stimulated (Experimental)
  Interventions: Device: Electric and electromagnetic stimulation

INTERVENTIONS:
Device: Electric and electromagnetic stimulation — Application of electromagnetic and electric stimulation using coils of different designs and electrodes to assess peripheral nerve sensitivity. The stimulation is momentary, non-therapeutic, and performed for basic science research purposes

SUMMARY:
Volunteers will undergo various peripheral nerve stimulations (electric, electromagnetic, and temporal interference) to evaluate each method's sensitivity. The main objective is to examine the relationship between nerve activation and coil placement relative to the nerve, as well as how different coil types influence maximal nerve activation.

ELIGIBILITY:
Inclusion Criteria:

* Person aged > 18 years
* Signed informed consent
* Healthy
* Willingness and ability to adhere to study procedures

Exclusion Criteria:

* Known hypersensitivity to electric or electromagnetic stimulation
* Any implanted metal or electronic device in the upper body (except dental work such as fillings or braces), e.g., active medical devices, metal implants
* Neurological or neuromuscular disorders or conditions
* History of seizures or epilepsy
* Current treatment with drugs that lower seizure threshold (e.g., certain analgesics, methylxanthines, antipsychotics, antidepressants, antiepileptics, anesthetics)
* Pregnancy or breastfeeding
* Surgical intervention of the arm within the last 4 weeks
* Allergy to adhesives or ultrasound gel components (e.g., polyethylene glycols)
* Skin lesions, infections, or strictures in the arm region
* Tattoos on the stimulated (right) arm and hand, or in any area likely to be captured in video recordings
* Inability to follow study procedures (e.g., due to language barrier, psychological disorders, dementia)
* Participant deprived of liberty by administrative or judicial decision or under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum nerve activation response to electromagnetic stimulation with different coils | Day 1
  Maximum of the measured signals (muscle contraction from electromyography (EMG) and finger movement from accelerometer) obtained across all stimulation positions at a given stimulation intensity for each coil type. This reflects the relative sensitivity of peripheral nerves to electromagnetic stimulation with different coil designs.

SECONDARY OUTCOMES:
Spatial range of nerve activation with electromagnetic coils | Day 1
  Distance around the stimulation position yielding the maximum response (E1), within which the measured signals (muscle contraction and finger movement) remain at least 50% of the maximum, across all coil positions at a given stimulation intensity.
Spatial range of nerve activation with neuromuscular electrical stimulation electrodes (NMES) | Day 1
  Distance around the stimulation position yielding the maximum response, within which the measured signals (muscle contraction and finger movement) remain at least 50% of the maximum, across all NMES electrode positions at a given stimulation intensity.
Amplitude ratios of temporal interference stimulation (TIS) electrodes associated with nerve activation | Day 1
  Electrode amplitude ratios during Temporal Interference Stimulation (TIS) for which measured signals remain at least 50% of the maximum signals observed at the optimal position.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Human Centered Engineering HuCE, Biel, Biel, Switzerland